CLINICAL TRIAL: NCT05613127
Title: A Randomized, Double-blind, Multicenter, Multinational, Active-controlled, Parallel-designed Phase 3 Clinical Trial to Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in Healthy Children Aged From 24months to 15yrs
Brief Title: To Evaluate the Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in Healthy Children Aged From 24mons-15yrs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boryung Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BR-HAV-CT-303
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis A; Hep A
Keywords: Hepatitis A; Hepatitis A vaccine; Vaccine; Hep A; HAV
MeSH Terms: conditions — Hepatitis A; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Inactivated Hepatitis A vaccine
  Interventions: Biological: Boryung Hepatitis A Vaccine Pre-Filled Syringe Inj. 0.5 mL
- Control group (Active Comparator): Inactivated Hepatitis A vaccine
  Interventions: Biological: HAVRIX 720 Junior 0.5 mL

INTERVENTIONS:
Biological: Boryung Hepatitis A Vaccine Pre-Filled Syringe Inj. 0.5 mL — Dosage and administration: pre-iflled syringe, IM injection of 0.5mL will be given for 2 times with 6-months interval.
  Arms: Test group
Biological: HAVRIX 720 Junior 0.5 mL — Dosage and administration: pre-filled syringe, IM injection of 0.5mL will be given for 2 times with 6-months interval.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate immunogenicity and safety of inactivated hepatitis A vaccine in healthy children aged from 24 months to 15 years when administered an initial dose followed by a booster dose (a total of 2 doses administered with 6 months interval).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate immunogenicity and safety of inactivated hepatitis A vaccine in healthy children aged from 24 months to 15 years when administered an initial dose followed by a booster dose (a total of 2 doses administered with 6 months interval).

This study is a two-group comparative study using a marketed inactivated hepatitis A vaccine (HAVRIX®, manufactured by GSK) as a control. The study will demonstrate non-inferiority of the test vaccine compared to the control vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female children ≥ 24 months and ≤ 15 years old on the day of first vaccination
2. Subjects with no history of hepatitis A and no previous vaccination against hepatitis A
3. Written informed consent obtained from the subject's legal representative (parents or representative)
4. Children who no health issues based on medical history and physical examination as judged by the investigator

Exclusion Criteria

1. Tympanic temperature of 38.0℃ or above within 48 hours prior to vaccination or on the day of vaccination
2. Uncontrolled epilepsy or neurological disorder
3. History of thrombocytopenia or has a risk of bleeding
4. History of hypersensitivity to the following: neomycin, formaldehyde, gentamicin sulfate, any vaccine
5. Severe acute or chronic infectious disease on the day of vaccination
6. Congenital / acquired immunodeficiency or receiving immunosuppressive therapy
7. Received immunosuppressive dose of systemic corticosteroids within 12 weeks prior to the first vaccination with the IP (Investigational Product) (equivalent potency of ≥ prednisolone 20 mg/day or equivalent potency of ≥ prednisolone 2.0 mg/kg/day in < 10kg of body weight for ≥ 14 consecutive days)
8. Administration of any other vaccine within 4 weeks prior to Screening
9. Planned administration of any other vaccine within 4 weeks after the last vaccination of the investigational product
10. Administration of immunoglobulins or blood products or received blood transfusion within 12 weeks prior to Screening
11. Currently participating in another clinical trial or administered / applied other investigational product / medical device within 6 months prior to Screening
12. Ineligibility for participate in the study for other reasons as determined by the investigator

Ages: 24 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Anti-HAV seroconversion rate at 4 weeks after the second vaccination | At Visit 6 (7 months after Day 1: first vaccination)
  Seroconversion: anti-HAV ≥ 20 mIU/mL after the second vaccination in subjects with anti-HAV < 20 mIU/mL at baseline

SECONDARY OUTCOMES:
GMCs (Geometric Mean Concentrations) measured with anti-HAV antibody titers at before the first vaccination and 4 weeks after the second vaccination | At Visit 6 (7 months after Day 1: first vaccination)
  GMCs (Geometric Mean Concentrations) measured with anti-HAV antibody titers at before the first vaccination and 4 weeks after the second vaccination
GMR (Geometric Mean Ratio, GMC Visit 6/GMC Visit 1) measured with anti-HAV antibody titers at 4 weeks after the second vaccination compared to those before the first vaccination | At Visit 6 (7 months after Day 1: first vaccination)
  GMR (Geometric Mean Ratio, GMC Visit 6/GMC Visit 1) measured with anti-HAV antibody titers at 4 weeks after the second vaccination compared to those before the first vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- The Catholic University of Korea, ST. Vincent's Hospital, Suwon, South Korea
- Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No